CLINICAL TRIAL: NCT01224860
Title: A Prospective, Randomized, Open Label Blinded End Point (Probe), Crossover Study to Compare the Effects of Telmisartan and Losartan on Metabolic Profile of Renal Transplant Patients
Brief Title: Telmisartan Versus Losartan in Kidney Transplantation
Acronym: COSTANT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: COSTANT; 2008-000822-38 (EudraCT Number)
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Renal Transplant
Keywords: Telmisartan; Losartan; Renal transplant
MeSH Terms: interventions — Telmisartan; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telmisartan (Experimental)
  Interventions: Drug: Telmisartan
- Losartan (Experimental)
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Telmisartan — One week 40 mg daily, followed by fifteen weeks treatment period with 80 mg daily.
  Arms: Telmisartan
Drug: Losartan — One week 50 mg daily, followed by fifteen weeks treatment period with 100 mg daily.
  Arms: Losartan

SUMMARY:
In renal transplant recipients, residual renal insufficiency combined to the effects of immunosuppressive therapy with steroids or calcineurin inhibitors may reduce insulin activity and may contribute to several of the abnormalities associated with the metabolic syndrome, such as hypertension, glucose intolerance and hyperlipidemia. In turn, insulin resistance, hypertension, hyperglycemia and dyslipidemia may importantly contribute to the excess cardiovascular risk of renal transplant patients (an excess comparable to that of diabetes subjects with over diabetic nephropathy)and may also accelerate progressive renal function deterioration and promote graft loss. Thus, amelioration of the insulin activity and of the related metabolic syndrome is a key component of treatments aimed to improve patient and graft survival in renal transplant recipients. Recently, drugs such as peroxisome proliferators-activated receptor-gamma activators, that ameliorate insulin sensitivity and metabolic syndrome, have become available.These agents, however, can provoke fluid retention, weight gain, edema and, in some cases, heart failure.

Recent studies showed that telmisartan, an angiotensin II type 1 receptor antagonist, in addition to block the angiotensin II type 1 - a key surface receptor involved in the regulation of blood pressure - may also activate peroxisome proliferators-activated receptor-gamma activators, thus improving some of the features of the metabolic syndrome. Thus telmisartan may substantially reduce the overall cardiovascular and renal risk of renal transplant recipients by ameliorating some of the modifiable components of the metabolic syndrome. On the other hand, telmisartan is devoid of the adverse effects of peroxisome proliferators-activated receptor-gamma activators such as fluid retention, and has therefore a remarkably better risk/benefit profile. Thus, whether telmisartan in addition to the beneficial effects of a reference angiotensin II type 1 receptor antagonist (such as losartan) may offer adjunctive advantages related to improved insulin sensitivity in renal transplant patients on chronic therapy with steroids and/or calcineurin inhibitors, is worth investigating.

DETAILED DESCRIPTION:
BACKGROUND In renal transplant recipients, residual renal insufficiency combined to the effects of immunosuppressive therapy with steroids or calcineurin inhibitors may reduce insulin activity and may contribute to several of the abnormalities associated with the metabolic syndrome, such as hypertension, glucose intolerance and hyperlipidemia. In turn, insulin resistance, hypertension, hyperglycemia and dyslipidemia may importantly contribute to the excess cardiovascular risk of renal transplant patients (an excess comparable to that of diabetes subjects with over diabetic nephropathy)and may also accelerate progressive renal function deterioration and promote graft loss. Thus, amelioration of the insulin activity and of the related metabolic syndrome is a key component of treatments aimed to improve patient and graft survival in renal transplant recipients. Recently, drugs such as peroxisome proliferators-activated receptor-gamma activators, that ameliorate insulin sensitivity and metabolic syndrome, have become available. These agents, however, can provoke fluid retention, weight gain, edema and, in some cases, heart failure. Thus, the risk/benefit profile of peroxisome proliferators-activated receptor-gamma activators is still uncertain, in particular in renal transplant patients where the risks of therapy may overwhelm the potential benefits.

Recent studies showed that telmisartan, an angiotensin II type 1 receptor antagonist, in addition to block the angiotensin II type 1 - a key surface receptor involved in the regulation of blood pressure - may also activate PPAR-gamma, thus improving some of the features of the metabolic syndrome, such as hyperglycemia and dyslipidemia in people with hypertension and/or diabetes. Thus, in addition to control high blood pressure and to limit some of the adverse effects of angiotensin II, including target organ damage, graft fibrosis and cyclosporine (CsA) nephrotoxicity, telmisartan may also substantially reduce the overall cardiovascular and renal risk of renal transplant recipients by ameliorating some of the modifiable components of the metabolic syndrome, such as hypertension, glucose intolerance and hyperlipidemia. On the other hand, telmisartan is devoid of the adverse effects of peroxisome proliferators-activated receptor-gamma activators such as fluid retention, and has therefore a remarkably better risk/benefit profile. Thus, whether telmisartan in addition to the beneficial effects of a reference AII receptor antagonist (such as losartan) may offer adjunctive advantages related to improved insulin sensitivity in renal transplant patients on chronic therapy with steroids and/or calcineurin inhibitors, is worth investigating.

AIMS The primary aim is to compare the short-term effects of telmisartan and losartan on insulin sensitivity in kidney transplant recipients with stable renal function and concomitant treatment with steroids and/or calcineurin inhibitors.

DESIGN This will be a pilot, explorative study. On the basis of previous experimental evidence, a crossover study on 20 patients should have the power to detect a statistically significant difference in the effect on insulin activity between each treatment period as compared to baseline.

Patients will be randomised on a 1:1 basis to the sequence Telmisartan-Losartan or to sequence losartan-telmisartan.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent;
* Age > 18 years;
* Single renal transplant or dual marginal > 6 months duration;
* Blood pressure >130/85 mmHg or need for anti-hypertensive therapy;
* Stable renal function (changes in serum creatinine < 30%) and no acute rejection episodes in the last six months;
* Stable (for at least six months) dual or triple immunosuppressive therapy including corticosteroids or calcineurin inhibitors;
* Legal capacity.

Exclusion Criteria:

* Vascular disease of the kidney;
* Heart failure: NYHA classification class III-IV on ACE or AII inhibitor therapy;
* Cerebral haemorrhage, stroke or TIA within three months prior to study enrolment;
* Myocardial infarction within three months prior to study enrolment;
* Unstable angina pectoris;
* Severe hepatic disease;
* Pregnancy or women of child-bearing potential without following a scientifically accepted form of contraception;
* Overt diabetes or concomitant treatment with oral antidiabetic agents and/or insulin;
* Specific clinical indication (other than arterial hypertension) to be treated with ACE inhibitors or AII receptor antagonists;
* Specific contraindications or history of hypersensitivity to the study drugs, glitazones, ACE inhibitors or AII receptor antagonists;
* Participation to other clinical trials over the last three months;
* Legal incapacity;
* Previous diagnosis of: intellectual disability/mental retardation, dementia, schizophrenia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity. | At baseline and then every four months.
  Glucose disposal rate as assessed by an euglycemic hyperinsulinemic clamp.
Insulin sensitivity. | At 9 month.
  Glucose disposal rate as assessed by an euglycemic hyperinsulinemic clamp.

SECONDARY OUTCOMES:
Systemic variables. | At baseline and then every four months.
  Sitting systolic/diastolic blood pressure, 24-h blood pressure profile.
Systemic variables. | At 9 month.
  Sitting systolic/diastolic blood pressure, 24-h blood pressure profile.
Metabolic variables. | At baseline and then every four months.
  Morning fasting blood glucose, Glucose tolerance test, Glicated hemoglobin, Morning fasting insulin, HOMA index, Lipid profile (total cholesterol, triglycerides, HDL, LDL, apolipoprotein A, B.
Metabolic variables. | At 9 month.
  Morning fasting blood glucose, Glucose tolerance test, Glicated hemoglobin, Morning fasting insulin, HOMA index, Lipid profile (total cholesterol, triglycerides, HDL, LDL, apolipoprotein A, B.
Renal variables. | At baseline and then every four months.
  UAE (as assessed by nephelometry in three consecutive overnight urine collections), GFR/RPF (as assessed by Iohexol and PAH plasma clearance, respectively), Albumin fractional clearance.
Renal variables. | At 9 month.
  UAE (as assessed by nephelometry in three consecutive overnight urine collections), GFR/RPF (as assessed by Iohexol and PAH plasma clearance, respectively), Albumin fractional clearance.

CONTACTS AND LOCATIONS:
Locations (1):
- Mario negri Institute - Clinical Research Center for Rare Diseases, Ranica, Bergamo, Italy

REFERENCES:
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471